CLINICAL TRIAL: NCT04894266
Title: An Open-Label Study to Assess the Safety and Effect on Clinical Course and Key Biomarkers of Oral Apabetalone in Hospitalized Subjects With Covid-19 Infection in Addition to Standard of Care (SOC)
Brief Title: An Open-Label Study of Apabetalone in Covid Infection
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unable to recruit subjects
Sponsor: Resverlogix Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RVX222-CS-023
Record Dates: First submitted 2021-05-05; First posted 2021-05-20 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — apabetalone; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is an open-label, exploratory clinical study to assess the patient safety and effect of oral apabetalone for up to 4 weeks in hospitalized subjects with Covid-19 infection. Subjects at each center will be randomized into 2 cohorts to receive SOC plus apabetalone or SOC alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other): All subjects will receive SOC during their hospital admission. This will include daily vital signs, WHO Ordinal Scale assessment and adverse events. On Days 3, 5, 7 and 11, hematology, chemistry, oropharyngeal or nasopharyngeal swabs for Covid-19 viral levels and biomarkers samples the same as at the screening visit will be taken if the patient remains in hospital.
  Interventions: Other: Standard of care
- Standard of Care plus apabetalone (Experimental): All subjects will receive SOC during their hospital admission. This will include daily vital signs, WHO Ordinal Scale assessment and adverse events. On Days 3, 5, 7 and 11, hematology, chemistry, oropharyngeal or nasopharyngeal swabs for Covid-19 viral levels and biomarkers samples the same as at the screening visit will be taken if the patient remains in hospital. For the apabetalone cohort, treatment will be administered BID with meals.
  Interventions: Drug: Apabetalone; Other: Standard of care

INTERVENTIONS:
Drug: Apabetalone — Apabetalone 100mg BID
  Arms: Standard of Care plus apabetalone
Other: Standard of care — Standard of Care

SUMMARY:
The primary objective of the study is to evaluate the safety and effect on clinical course of oral apabetalone in hospitalized subjects with Covid-19 infection

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of the study is to evaluate the safety and effect on clinical course of oral apabetalone in hospitalized subjects with Covid-19 infection

Secondary Objectives:

To evaluate the effect of apabetalone on biomarkers of inflammation (interleukin [IL]-6, IL-8, tumor necrosis factor [TNF]-α and C-reactive protein [CRP]) To evaluate the effect of apabetalone on key virus-related biomarkers including ACE2, serine protease inhibitor Clade A Member 8 (SERPINA8), angiotension (Ang) II and Ang (1-7) and others within the renin-angiotensin system (RAS) To evaluate the effect of apabetalone on clinical laboratory parameters including white blood cell (WBC) count, platelet count, D-Dimer, ferritin and clotting time in hospitalized subjects with Covid-19 infection To evaluate the effect of apabetalone cardiac and renal biomarkers including N-terminal pro B-type natriuretic peptide (NT-proBNP), troponin and Cystatin C To evaluate changes in viral levels measured via oropharyngeal or nasopharyngeal swabs To evaluate the effect of apabetalone on rate of admission to ICU, need for mechanical ventilation/ECMO, and death To evaluate the safety of apabetalone in hospitalized subjects with Covid-19 Infection

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent before participation in the study.
2. Aged ≥18 years
3. Hospital admission with symptoms suggestive of COVID-19 infection
4. Ten days or less since the onset of symptoms
5. Virological confirmation of SARS-CoV2 infection by reverse transcriptase PCR (RT- PCR) according to Center for Disease Control and Prevention (CDC) guidelines within the previous 72 hours
6. Subjects showing bilateral pulmonary infiltrates on chest imaging
7. Saturation of oxygen (SpO2) by pulse oximetry <94% on room air at sea level.
8. Female subjects must meet one of the following:

   * If of childbearing potential, female subjects must have a negative urine pregnancy test at screening and must also be willing to practice total abstinence or to use an approved (non-hormonal) form of birth-control throughout the study treatment phase and up to 28 days after the last study drug dose if randomized to apabetalone." -OR-
   * Meet at least one of the following criteria:
   * Be postmenopausal, defined as having been amenorrheic for at least 2 years
   * Have had a hysterectomy or a bilateral oophorectomy

Exclusion Criteria:

1. Subjects with SpO2 >94% on room air using pulse oximetry and without bilateral infiltrates on chest imaging
2. Subjects requiring mechanical ventilation or extracorporeal membrane oxygenation
3. Patients with Stage 5 CKD receiving renal replacement therapy with either hemodialysis or peritoneal dialysis, renal transplant or with eGFR <15 mL/min/1.73 m2.
4. Patients with prior transplantations of organs or bone marrow.
5. Patients with unstable cardiac condition including heart attack, stroke, uncontrolled atrial fibrillation or a major cardiac procedure within 3 months as assessed by the investigator.
6. New York Heart Association Class IV congestive heart failure.
7. Evidence of cirrhosis from liver imaging or biopsy, a history of hepatic encephalopathy, esophageal or gastric varices, active hepatitis, or prior porta-caval shunt procedure.
8. ALT or AST >5 x ULN on admission laboratory assessment.
9. Total bilirubin >2 x ULN on admission laboratory assessment.
10. Have received any live attenuated vaccine within 90 days at dosing.
11. Known human immunodeficiency virus positive patients.
12. Chronic use of oxygen therapy at home
13. Have participated in a clinical study and received any investigational medication within the last 30 days preceding Visit 1 (Screening).
14. Subjects whose safety may be compromised by study participation
15. Are not, in the opinion of the investigator, able or willing to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the change in WHO Ordinal Scale for Clinical Improvement at Day 14 | Change in WHO Ordinal Scale for Clinical Improvement at Day 14
  WHO Ordinal Scale for Clinical Improvement, 8 point scale, 0 = no clinical or virological evidence of infection

SECONDARY OUTCOMES:
Change in WHO Ordinal Scale for Clinical Improvement at Day 28 | Study Day 28
  WHO Ordinal Scale for Clinical Improvement, 8 point scale, 0 = no clinical or virological evidence of infection
Biomarkers of inflammation Interleukin-6 | Study Day 28
  Interleukin-6 is a biomarker of inflammation
Total time of hospitalization | through study completion, an average of 28 days
  Total time of hospitalization
Biomarkers of inflammation Interleukin-8 | Study Day 28
  Interleukin-8 is a biomarker of inflammation
Biomarkers of inflammation Tumor Necrosis Factor alpha | Study Day 28
  Tumor Necrosis Factor alpha is a biomarker of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No